CLINICAL TRIAL: NCT02555124
Title: A Double-Blind, Placebo-Controlled, Randomized, Single-Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of JNJ-42847922 in Healthy Japanese Male Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of JNJ-42847922 in Healthy Japanese Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107878; 42847922ISM1002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2015-09-18; First posted 2015-09-21 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: Healthy; JNJ-42847922
MeSH Terms: interventions — seltorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A (Experimental): Participants will receive single oral dose of 5 milligram (mg) of JNJ-42847922 or Placebo on Day 1, fasted condition.
  Interventions: Drug: JNJ-42847922, 5 mg; Drug: Placebo
- Cohort B (Experimental): Participants will receive single oral dose of 20 mg of JNJ-42847922 or Placebo on Day 1, fasted condition.
  Interventions: Drug: JNJ-42847922, 20 mg; Drug: Placebo
- Cohort C (Experimental): Participants will receive single oral dose of 40 mg of JNJ-42847922 or Placebo on Day 1, fasted condition.
  Interventions: Drug: JNJ-42847922, 40 mg; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42847922, 5 mg — Participants will receive single oral dose of 5 milligram (mg) of JNJ-42847922 on Day 1, fasted condition.
  Arms: Cohort A
Drug: JNJ-42847922, 20 mg — Participants will receive single oral dose of 20 mg of JNJ-42847922 on Day 1, fasted condition.
  Arms: Cohort B
Drug: JNJ-42847922, 40 mg — Participants will receive single oral dose of 40 mg of JNJ-42847922 on Day 1, fasted condition.
  Arms: Cohort C
Drug: Placebo — Participants will receive placebo on Day 1, fasted condition in Cohort A, Cohort B and Cohort C.

SUMMARY:
The purpose of this study is to evaluate the safety of JNJ-42847922 following single oral administration.

DETAILED DESCRIPTION:
This is a single center, double-blind (neither the researchers nor the participants know what treatment the participant is receiving), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect), randomized (study medication assigned to participants by chance), single-ascending dose study. The study consists of a screening phase, an in-clinic treatment phase, and a follow-up phase. The study duration for each subject will be approximately 5 weeks from screening (Day -28 to Day -3), in-clinic period (Day -2 to Day 4) to follow up visit (Day 8). Participants will receive a single oral dose of JNJ-42847922 or placebo in 3 cohorts. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be willing and able to adhere to the prohibitions and restrictions specified inprotocol, Prohibitions and Restrictions
* A man who is sexually active with a woman of childbearing potential and has not had avasectomy must agree to use an adequate contraception method as deemed appropriate by the investigator (eg, vasectomy, double-barrier, partner using effective contraception), and all men must also agree not to donate sperm during the study and for 3 months afterreceiving the last dose of study drug
* Participant must have a body mass index (BMI) between 18.0 and 29.9 kilogram per square meter (kg/m^2), and body weight not less than 50 kg
* Participant must have a 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function, Including: Synus rhythm; Heart rate between 45 and 99 beats per minute (bpm); QT corrected according to Fridericia's formula (QTcF) interval less than or equal to (<=)450 milliseconds (ms); QRS interval of <=120 ms; PR interval <=220 ms; Morphology consistent with healthy cardiac conduction and function
* Nonsmoker (not smoked for 3 months prior to screening)

Exclusion Criteria:

* Participant has a history of or current clinically significant medical illness including (but notlimited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulationdisorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities,significant pulmonary disease, including bronchospastic respiratory disease, diabetesmellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease,infection, or any other illness that the investigator considers should exclude the participant orthat could interfere with the interpretation of the study results
* Participant has a clinically significant abnormal value for hematology, coagulation,biochemistry, or urinalysis at screening as deemed appropriate by the investigator
* Participant has a clinically significant abnormal physical examination, neurologic examination,or vital signs as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbalsupplements), except for acetaminophen within 14 days before study drug administration onDay 1
* Participant has known allergies, hypersensitivity, or intolerance to JNJ-42847922 or its excipients

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09-12 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | up to Day 8
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of Participants With Serious Adverse Events (SAEs) | up to Day 8
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Day 1 (pre-dose), 0.16, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,16 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48, 60 hr post-dose on Day 3; 72 hr post-dose on Day 4
  Cmax is the maximum observed plasma concentration.
Time to Reach the Maximum Observed Plasma Concentration (Tmax) | Day 1 (pre-dose), 0.16, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,16 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48, 60 hr post-dose on Day 3; 72 hr post-dose on Day 4
  Tmax is the time to reach the maximum observed plasma concentration.
Time to Last Time of the Last Measurable (nonbelow quantification limit [nonBQL]) Plasma Concentration (Tlast) | Day 1 (pre-dose), 0.16, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,16 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48, 60 hr post-dose on Day 3; 72 hr post-dose on Day 4
  Tlast is the time to last time of the last measurable (nonbelow quantification limit [nonBQL]) plasma concentration.
AUC From Time 0 to the Time of the Last Measurable (nonBQL) Plasma Concentration (AUClast) | Day 1 (pre-dose), 0.16, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,16 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48, 60 hr post-dose on Day 3; 72 hr post-dose on Day 4
  AUClast is the area under the plasma concentraion curve from time 0 to the time of the last measurable (nonBQL) plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Day 1 (pre-dose), 0.16, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,16 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48, 60 hr post-dose on Day 3; 72 hr post-dose on Day 4
  The AUC(0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Percentage of Area Under the Plasma Concentrationtime Curve Obtained by Extrapolation (%AUC [infinity,ex]) | Day 1 (pre-dose), 0.16, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,16 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48, 60 hr post-dose on Day 3; 72 hr post-dose on Day 4
  Percentage of area under the plasma concentration-time curve obtained by extrapolation (%AUC[inf,ex]) is calculated by dividing the difference of AUC(0-infinity) and AUC(0-last) by AUC(0-infinity) and then multiplying by 100 (AUC[0-infinity] - AUC[0-last])*100/AUC[0-infinity].
Apparent Elimination Half-life (t1/2) | Day 1 (pre-dose), 0.16, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,16 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48, 60 hr post-dose on Day 3; 72 hr post-dose on Day 4
  Elimination half-life (t [1/2]) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Apparent Terminal Elimination Rate Constant (Lambda[z]) | Day 1 (pre-dose), 0.16, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,16 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48, 60 hr post-dose on Day 3; 72 hr post-dose on Day 4
  Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Total Apparent Clearance (CL/F) | Day 1 (pre-dose), 0.16, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,16 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48, 60 hr post-dose on Day 3; 72 hr post-dose on Day 4
  Total apparent clearence is calculated as dose divided by AUC(infinity).
Apparent Volume of Distribution (Vd/F) | Day 1 (pre-dose), 0.16, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,16 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48, 60 hr post-dose on Day 3; 72 hr post-dose on Day 4
  Apparent volume of distribution is calculated as Dose divided by Lambda[z] multiplied by AUC(infinity).
Change From Baseline in Stanford Sleepiness Scale Score at Day 1 | Baseline and Day 1
  The Stanford Sleepiness Scale (SSS) is a subjective rating of sleepiness, with score ranging from 1 to 7, where higher values reflect more severe sleepiness

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Osaka, Japan